CLINICAL TRIAL: NCT03396731
Title: A Prospective, Multicentre, Randomised, Assessor Blinded Study Comparing the Efficacy, Including Patient Reported Outcomes of Two Different Daily gekoTM Treatment Durations in Conjunction With Standard Care, With Each Other and to Standard Care Alone, in Patients With Venous Leg Ulcers
Brief Title: Efficacy Study for Geko Device in VLU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSK-VLU-004
Record Dates: First submitted 2017-09-12; First posted 2018-01-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Venous Leg Ulcer; Leg Ulcers Venous; Leg Ulcer; Wound Leg; Wound
Keywords: VLU; Venous Leg Ulcer; Leg Ulcer; Leg Wound
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors will be blinded to the study participants and what treatment they are receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care alone (control) (No Intervention): Multilayer/multi component compression bandaging treatment
- 6 hours geko™ (no longer recruiting) (Active Comparator): geko™ device 6 hours daily for 4 weeks treatment phase, to be used in conjunction with Standard of care.
  Interventions: Device: geko™ medical device
- 12 hours geko™ (Active Comparator): geko™ device 12 hours daily for 4 weeks treatment phase, to be used in conjunction with Standard of care.
  Interventions: Device: geko™ medical device

INTERVENTIONS:
Device: geko™ medical device — The geko™ device, manufactured by Firstkind Ltd (High Wycombe, United Kingdom), is a small disposable, battery powered CE marked medical device.
  Arms: 12 hours geko™; 6 hours geko™ (no longer recruiting)

SUMMARY:
Eight weeks, comprised of four weeks Run-in Phase of Standard Care (SC) treatment followed by four weeks of treatment allocated by randomisation (Treatment Phase).

To compare two daily geko™ device treatment durations, six hours and 12 hours, in conjunction with SC, with each other and to SC alone, in patients with venous leg ulcers

DETAILED DESCRIPTION:
1. Screen patient database to identify eligible patients
2. Obtain informed consent and inform participant's GP
3. Complete CRF throughout the study period (demographics, vital signs, medical history, study ulcer history, concomitant medication)
4. Physical examination at the study start up visit and at consecutive weekly visits
5. Take a digital image of the wound at participants weekly visits
6. Assess and report adverse events
7. Apply standard care (compression bandaging) at weekly visits and record all the dressing usage
8. Perform randomisation at the end of week 4 and allocate participant to one of the three treatment groups.
9. Train the participant to use gekoTM devices
10. Schedule weekly visits

ELIGIBILITY:
Inclusion Criteria:

Potential subjects are required to meet all of the following criteria for enrollment into the study and subsequent randomization.

1. Male or female aged ≥ 18 years and able to provide written informed consent.
2. Intact healthy skin at the site of gekoTM device application.
3. Patients who have a chronic venous leg ulcer determined to be due to underlying venous disease following evaluation in a multidisciplinary clinic setting.
4. A VLU of approximately ≥ 3cm2 and ≤ 39 cm2 at study enrolment i.e. Run In Phase Visit 1 (RV1). The largest ulcer within the given size range will be designated the study ulcer and the only one included in the study. If other ulcerations are present on the same leg they have to be more than 2 cm apart if they are separate wounds.
5. Study ulcer (current episode of ulceration in case of ulcer recurrence) has been present for at least 6 weeks but no more than 5 years prior to study entry (i.e. RV1).
6. Ankle-Brachial Pressure Index (ABPI) of 0.75-1.24 inclusive measured at study entry or within 8 weeks prior to study entry (i.e. RV1).
7. No active local or systemic infection for a minimum of 48 hours prior to study entry (i.e. RV1).
8. No systemic antimicrobial treatment for a minimum of seven days prior to study entry prescribed for index wound infection (i.e. RV1).
9. Patient understands and is willing to participate in the study and is able to comply with study procedures and visits.

Note: At the randomisation visit, the study ulcer needs to be ≥ 2 cm2 and ≤ 30 cm2.

Exclusion Criteria:

Potential subjects meeting any of the following criteria will be excluded from enrollment and subsequent randomisation:

1. Known allergy to any of the protocol-stipulated treatments, or non-tolerance of multilayer, multicomponent compression therapy.
2. History of significant haematological disorders (e.g. Sickle Cell disease).
3. History of Deep Vein Thrombosis (DVT) within six months preceding study entry (i.e. RV1).
4. History of Pyoderma Gangrenosum or other inflammatory ulceration.
5. Pregnancy or breast feeding.
6. Use of investigational drug or device within four weeks prior to study entry (i.e. RV1) that may interfere with this study.
7. Use of any neuro-modulation device.
8. Surgery during three months prior to study entry (such as abdominal, gynaecological, hip or knee replacement) (i.e. RV1).
9. Trauma to the lower limbs that would prevent geko™ from stimulating the common peroneal nerve.
10. No involuntary movement of the lower leg/foot at the maximum tolerable device setting.
11. Any medication deemed by the Investigator to potentially interfere with the study treatment (e.g. systemic steroids).
12. Participation in any other clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Linear healing rate (LHR) | 8 weeks
  Linear healing rate will be studied on a weekly basis

SECONDARY OUTCOMES:
Wound healing rate | Upto 8 weeks
  Measured with the images taken
Pain reduction | Upto 8 weeks
  Participant reported outcome of pain reduction using Visual Analogue Scale (VAS)
Change in Quality of Life | Upto 8 weeks
  Change in Quality of Life based on participant reported outcomes using EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Keith Harding, FRCGP FRCP FRCS, Principal Investigator — Welsh Wound Innovation Centre
Locations (23):
- United Kingdom (23):
  - Trafalgar Group Medical Practice, Southsea, Portsmouth
  - Crouch Oak Family Practice, Addlestone
  - Barnsley Hospital NHS foundation Trust, Barnsley
  - Heart of Bath Medical Partnership, Bath
  - West Walk Surgery, Bristol
  - Rowden Surgery, Chippenham
  - Lakeside Healthcare, Corby
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - South Tyneside NHS Foundation Trust, Hebburn
  - The Queen Elizabeth Hospital King's Lynn NHS Foundation Trust, Kings Lynn
  - Lancashire Care NHS Trust, Leyland
  - Accelerate CIC, London
  - Royal Free London NHS Foundation Trust, London
  - Central London Community Healthcare, London
  - Norfolk Community Health and Care NHS Trust, Norwich
  - Norfolk and Norwich University Hospital, Norwich
  - The Adam Practice, Poole
  - Hertfordshire Community NHS Trust, Stevenage
  - Musgrove Park Hospital, Taunton
  - Breckland Alliance, Thetford
  - Welsh wound Innovation Centre, Wales
  - Worcestershire Royal Hospital, Worcester
  - York Teaching Hospital NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bull RH, Clements D, Collarte AJ, Harding KG. The impact of a new intervention for venous leg ulcers: A within-patient controlled trial. Int Wound J. 2023 Aug;20(6):2260-2268. doi: 10.1111/iwj.14107. Epub 2023 Feb 13. PMID 36785909
- [Result] Bull RH, Clements D, Collarte AJ, Harding KG. A Novel Randomized Trial Protocol for Evaluating Wound Healing Interventions. Adv Wound Care (New Rochelle). 2023 Dec;12(12):671-679. doi: 10.1089/wound.2023.0058. Epub 2023 Sep 5. PMID 37526355
- See also: Device official website — http://www.gekodevices.com/en-uk/
- See also: Publication- International Wound Journal — http://www.onlinelibrary.wiley.com/doi/10.1111/iwj.14107

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03396731/Prot_SAP_000.pdf